CLINICAL TRIAL: NCT02227160
Title: Group Interventions for Suicidal African Americans
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study never started enrolling participants due to lack of grant funding.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nadine Kaslow, PhD, Nadine Kaslow PhD, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00073021
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Depression; Mental Illness; Suicide; Suicidal Ideation
MeSH Terms: conditions — Depression; Mental Disorders; Suicide; Suicidal Ideation | interventions — Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychosocial group intervention (Experimental): Subjects will seek outpatient counseling, support groups, in addition to 10 weekly group meetings
  Interventions: Behavioral: 10 weekly group meetings; Behavioral: Outpatient counseling and support groups
- Control (Active Comparator): Subjects will seek outpatient counseling and support groups only
  Interventions: Behavioral: Outpatient counseling and support groups

INTERVENTIONS:
Behavioral: 10 weekly group meetings — 10 weekly group meetings with up to five other men and women at Grady Health System
  Arms: Psychosocial group intervention
Behavioral: Outpatient counseling and support groups — Usual mental health care

SUMMARY:
The investigator is conducting a hybrid efficacy-effectiveness randomized controlled trial with low-income African American suicide attempters. Guided by the Theory of Triadic Influence (TTI), this pilot randomized controlled trial aims:

1. to determine if psychosocial group intervention (PGI) is more effective than enhanced treatment as usual (ETAU) in reducing suicidal behavior (ideation, attempts; primary outcome) and improving its correlates (depressive symptoms, hopelessness, quality of life) (secondary outcomes) in low-income African Americans with a recent attempt.
2. to determine if PGI is more effective than ETAU at bolstering intrapersonal (I), social/situational (SS), and cultural/environmental (CE) risk and protective factors that mediate the condition-suicidal behavior and correlates link and thus serve as mechanisms of change.
3. to determine I, SS, and CE variables that moderate the condition-suicidal behavior link and thus serve as predictors of intervention outcome.

Hypothesis for Aim 1: At post-intervention and follow-up, PGI participants will evidence greater improvements in suicidal behavior and its correlates than those in ETAU.

Hypothesis for Aim 2: Changes in these risk and protective factors will account for condition effects on outcomes: (1) psychological distress, aggression, impulsivity, substance abuse, low self-esteem, and suicide acceptability (I-risk); (2) perceived burdensomeness and thwarted belongingness, relationship discord, intimate partner violence perpetration and victimization (SS-risk); (3) access to a weapon and barriers to service utilization (CE-risk); (4) reasons for living, optimism, positive ethnic identity, effective coping, and spiritual well-being (I-protective); (5) overall family health and social support from family and friends (SS-protective); and (6) religious involvement and effectiveness of obtaining resources (CE-protective).

Hypothesis for Aim 3: Individuals (1) having fewer Diagnostic and Statistical Manual of Mental Disorders (DSM) disorders and attachment styles characterized by positivity toward the self and others (I); (2) children and more limited trauma histories (SS); and (3) more daily hassles and less exposure to community disorder (CE) will evidence greater reductions in suicidal behavior and its correlates and greater enhancements in quality of life at post-intervention and follow-up.

DETAILED DESCRIPTION:
Attention will be paid to Theory of Triadic Influence intrapersonal, social/ situational, and cultural/ environmental risk and protective factors that impact outcomes. The central hypothesis is that compared to enhanced treatment as usual, through targeting Theory of Triadic Influence-risk and protective factors the culturally-informed, Theory of Triadic Influence-driven, empowerment based psychosocial group intervention will more positively alter trajectories in suicidal behaviors and its correlates. The rationale is that upon study completion, if data support the psychosocial group intervention value, they will facilitate our long-term goal of disseminating evidence-based culturally-relevant interventions.

In order to test the hypothesis that at post-intervention and 6 and 12-month follow-up, compared to individuals in ETAU, those in the PGI will endorse less I, SS, and CE risk factors, reduced suicidal ideation, depressive symptoms, and hopelessness, and greater levels of I, SS, and CE protective factors as well as increased quality of life, the study procedures will be as follows: Male and female participants between the ages of 18-64 will be recruited in the medical and psychiatric emergency rooms at GHS. Once the individual has been medically cleared and has provided informed consent, he/she will be screened for study appropriateness by trained project team members (10-20 minutes). If he/she meets inclusion criteria, study participation will include a 3-hour interview. All study measures will be read to each participant. Measures will assess background variables, suicidal behavior, depressive symptoms, hopelessness, quality of life, and I, SS, and CE risk and protective factors. All measures are psychometrically sound and appropriate for use with an African American population. Once the interview is over, the participant will be randomly assigned to either the PGI (10 group therapy sessions) or the ETAU condition (participation in a support group focused on suicidal behaviors plus suicidal behavior monitoring and help with accessing resources). The PGI, conducted in accord with the culturally informed, TTI-guided, and empowerment based group protocol, and the support group will be unstructured; both groups will last 120 minutes. Following the completion of the PGI or ETAU condition, the individuals will be assessed at post-intervention (3 hours), and at 6 month and 12 month follow-ups (3 hours each). To increase retention and reduce suicide risk, reminder phone calls will be made and texts sent on Relieflink, a suicide prevention app that received 1st prize in an App Challenge sponsored by Substance Abuse and Mental Health Services Administration.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 64 yrs old
* patients who seek treatment at Grady Health System (GHS) after a suicide attempt
* African American
* speak English

Exclusion Criteria:

* cognitive impairments
* medical instability

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change in scores on Beck Scale for Suicidal Ideation | Baseline, post-therapy, 6 months and 12 months after therapy
  Beck Scale for Suicidal Ideation is a 21-item instrumentation used to measure the current intensity of patients' specific attitudes, behaviors and plans to commit suicide.

SECONDARY OUTCOMES:
Change in scores on Beck Depression Inventory - II | Baseline, post-therapy, 6 months and 12 months after therapy
  Beck Depression Inventory - II is a 21-item, self-reported questionnaire used to assess characteristics of depression.
Change in scores on Beck Hopelessness Scale | Baseline, post-therapy, 6 months and 12 months after therapy
  Beck Hopelessness Scale is a 20-item true-false self-report scale that measures the level of negative expectations about the future held by respondents
Change in scores on WHO Quality of Life Brief Instrument | Baseline, post-therapy, 6 months and 12 months after therapy
  The WHOQOL-BREF instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment.
Patient Satisfaction | 12 months
  Intervention Satisfaction Survey (ISS)

OTHER OUTCOMES:
Change in the Symptom Checklist 90-Revised (SCL 90-R) scale | Baseline, post-therapy, 6 months and 12 months after therapy
  Symptom Checklist 90-Revised (SCL 90-R) questionnaire measures overall levels of psychological and physical functioning.
Change in scores for Alcohol Use Disorders Identification Test | Baseline, post-therapy, 6 months and 12 months after therapy
  Alcohol Use Disorders Identification Test (AUDIT) is a 10 question test to determine if a person's alcohol consumption may be harmful
Change in scores on Drug Abuse Screening Test | Baseline, post-therapy, 6 months and 12 months after therapy
  Drug Abuse Screening Test (DAST) is a 28-item self-report scale that is used as a screening instrument for the abuse of drugs other than alcohol.
Change in scores on Rosenberg Self-Esteem Scale (RSE) | Baseline, post-therapy, 6 months and 12 months after therapy
  A 10-item scale that measures global self-worth by measuring both positive and negative feelings about the self.
Changes in scores on Short Form Buss-Perry Aggression Questionnaire | Baseline, post-therapy, 6 months and 12 months after therapy
  Short Form Buss-Perry Aggression Questionnaire is a 12-item short form that assesses four aspects of aggressive behavior: physical aggression, verbal aggression, anger and hostility.
Changes in scores on Barratt Impulsiveness Scale | Baseline, post-therapy, 6 months and 12 months after therapy
  Barratt Impulsiveness Scale is a 30-item self-report questionnaire designed to assess general impulsiveness taking into account the multifactorial nature of the construct.
Change in scores on Suicide Acceptability Scale | Baseline, post-therapy, 6 months and 12 months after therapy
  Suicide Acceptability Scale is an 8-item measure of suicide acceptability
Changes in scores on Interpersonal Needs Questionnaire (INQ) | Baseline, post-therapy, 6 months and 12 months after therapy
  Interpersonal Needs Questionnaire (INQ) is a 15-item self-report measure of the constructs of thwarted belongingness and perceived burdensomeness as defined by the Interpersonal Theory of Suicide.
Change in scores on Dyadic Adjustment Scale | Baseline, post-therapy, 6 months and 12 months after therapy
  Dyadic Adjustment Scale is a 32-item self-report tool used to assess couple satisfaction and to evaluate how each partner within the couple perceives his or her relationship
Change in scores on Conflict Tactics Scale-Revised | Baseline, post-therapy, 6 months and 12 months after therapy
  Conflict Tactics Scale-Revised (CTS-2) is 78-item, self-administered questionnaire that assesses both positive and negative behaviors used in response to conflict between romantic partners in the past year
Clinical Demographic Questionnaire | Baseline
  Demographic questionnaire assesses demographic information as well as information regarding to access to weapons
Change in scores on Reasons for Living Inventory | Baseline, post-therapy, 6 months and 12 months after therapy
  Reasons for Living Inventory contains 12 possible reasons for living, which respondents rate regarding the importance each item would be for living if suicide were contemplated.
Change in scores on Life Orientation Test - Revised | Baseline, post-therapy, 6 months and 12 months after therapy
  Life Orientation Test - Revised is a 10-item test assessing generalized positive outcome expectancies
Change in scores on Multi-dimensional Inventory of Black Identity | Baseline, post-therapy, 6 months and 12 months after therapy
  The Multi-dimensional Inventory of Black Identity is designed to assess the three cross-situationally stable dimensions (Centrality, Regard, and Ideology)
Change in scores on Ways of Coping (Revised) Questionnaire | Baseline, post-therapy, 6 months and 12 months after therapy
  Ways of Coping (Revised) is self-reported questionnaire used to assess adaptive and maladaptive ways to cope with negative emotions or problematic situations
Change in scores on Africultural Coping Systems Inventory | Baseline, post-therapy, 6 months and 12 months after therapy
  Africultural Coping Systems Inventory is a 30-item measure of the culture-specific coping strategies used by African Americans in stressful situations and is grounded in an African-centered conceptual framework
Change in scores on Barriers to Accessing Services Scale | Baseline, post-therapy, 6 months and 12 months after therapy
Change in scores on Spiritual Well-Being Scale | Baseline, post-therapy, 6 months and 12 months after therapy
  Spiritual Well-Being Scale is a 20-item scale used for the assessment of both individual and congregational spiritual well-being
Change in scores on Family Assessment Device | Baseline, post-therapy, 6 months and 12 months after therapy
  Family Assessment Device is a 53 item questionnaire designed to evaluate families.
Change in scores on Social Support Behaviors Scale | Baseline, post-therapy, 6 months and 12 months after therapy
  Social Support Behaviors Scale is designed to assess supportive behavior available from family and from friends.
Changes in scores on Multidimensional Measure of Religious Involvement for African Americans | Baseline, post-therapy, 6 months and 12 months after therapy
  Multidimensional Measure of Religious Involvement for African Americans is a 12-item scale measuring religious indicators.
Change in score on Effectiveness of Obtaining Resources questionnaire | Baseline, post-therapy, 6 months and 12 months after therapy
Change in evaluation on Structured Clinical Interview for DSM-5-Research Version | Baseline, post-therapy, 6 months and 12 months after therapy
  Structured Clinical Interview for DSM-5-Research Version is semi-structured interview that allows researchers to make clinical diagnoses according to DSM criteria
Change in evaluation on Structured Clinical Interview for DSM-PD | Baseline, post-therapy, 6 months and 12 months after therapy
  The Structured Clinical Interview for DSM-PD is a semi-structured interview for making DSM-IV Axis II: Personality Disorder diagnoses
Change in scores on Relationship Scales Questionnaire | Baseline, post-therapy, 6 months and 12 months after therapy
  Relationship Scales Questionnaire is a scale that consists of 17 items to assess attachment patterns.
Change in scores on Childhood Trauma Questionnaire - Short Form (CTQ-SF) | Baseline, post-therapy, 6 months and 12 months after therapy
  The CTQ-SF is a 28-item self-report instrument for adults and adolescents that assesses retrospective child abuse and neglect
Change in scores on Survey of Recent Life Experiences scale | Baseline, post-therapy, 6 months and 12 months after therapy
  Survey of Recent Life Experiences is a 51-item self-report instrument that measures hassles for adults
Change in scores on Community Disorder Scale | Baseline, post-therapy, 6 months and 12 months after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Kaslow, PhD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617